CLINICAL TRIAL: NCT06886503
Title: Inspiratory Muscle Warm-up Improves 400-meter Performance in Elite Runners - Randomized Crossover Trial
Brief Title: Effects of Inspiratory Muscle Warm-up on Respiratory Variables, Physiological Indices, and 400-meter Performance in Elite Male Runners - Randomized Crossover Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Sport - National Research Institute, Poland (Other)
Collaborators: Hitit University, Corum, Turkey (Unknown)
Responsible Party: Principal Investigator, Tomasz Kowalski, Supervisor-Consultant, Institute of Sport - National Research Institute, Poland
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HI:2024-148
Record Dates: First submitted 2025-03-09; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Athletic Performance
Keywords: inspiratory muscle warm-up; running performance
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- IW-SHAM (Experimental): Inspiratory Muscle Warm-up Protocols In addition to athletic warm-up an athletic warm-up protocol, participants performed inspiratory muscle warm-up (IMW) using the POWERbreathe® Plus Blue Medium Resistance (POWERbreathe International Ltd., Warwickshire, England UK). In the sham arm, inspiratory muscle warm-up was performed at 15% of maximal inspiratory pressure (MIP). Each protocol consisted of two sets of 30 repetitions (Marostegan et al., 2022; Demirkan et al., 2025).
  Interventions: Other: Sham
- Inspiratory Warm-Up 40% MIP (Other): In addition to athletic warm-up an athletic warm-up protocol, participants performed inspiratory muscle warm-up (IMW) using the POWERbreathe® Plus Blue Medium Resistance (POWERbreathe International Ltd., Warwickshire, England UK). In the sham arm, inspiratory muscle warm-up was performed at 40% of maximal inspiratory pressure (MIP). Each protocol consisted of two sets of 30 repetitions (Marostegan et al., 2022; Demirkan et al., 2025).
  Interventions: Other: Inspiratory Warm-up - 40% MIP
- Inspiratory Warm-Up 60% MIP (Other): In addition to athletic warm-up an athletic warm-up protocol, participants performed inspiratory muscle warm-up (IMW) using the POWERbreathe® Plus Blue Medium Resistance (POWERbreathe International Ltd., Warwickshire, England UK). In the sham arm, inspiratory muscle warm-up was performed at 60% of maximal inspiratory pressure (MIP). Each protocol consisted of two sets of 30 repetitions (Marostegan et al., 2022; Demirkan et al., 2025).
  Interventions: Other: Inspiratory Warm-Up - 60% MIP
- Athletic Warm-up Only (Other): The athletic warm-up (AWU) consisted of 15 minutes of low-intensity running (rate of perceived effort 2-4 on 1-10 Borg Scale), followed by dynamic stretching exercises targeting the upper and lower extremities. In the final phase, running drills were performed, including three progressively increasing sprint efforts over a distance of approximately 30 meters.
  Interventions: Other: Inspiratory Warm-Up - 60% MIP; Other: Inspiratory Warm-up - 40% MIP; Other: Sham

INTERVENTIONS:
Other: Inspiratory Warm-Up - 60% MIP — Inspiratory Muscle Warm-up Protocols In addition to athletic warm-up an athletic warm-up protocol, participants performed inspiratory muscle warm-up (IMW) using the POWERbreathe® Plus Blue Medium Resistance (POWERbreathe International Ltd., Warwickshire, England UK). In the IW60 arm, inspiratory muscle warm-up was performed at 60% of maximal inspiratory pressure (MIP). Each protocol consisted of two sets of 30 repetitions (Marostegan et al., 2022; Demirkan et al., 2025).
  Arms: Athletic Warm-up Only; Inspiratory Warm-Up 60% MIP
Other: Inspiratory Warm-up - 40% MIP — Inspiratory Muscle Warm-up Protocols In addition to athletic warm-up an athletic warm-up protocol, participants performed inspiratory muscle warm-up (IMW) using the POWERbreathe® Plus Blue Medium Resistance (POWERbreathe International Ltd., Warwickshire, England UK). In the IW40 arm, inspiratory muscle warm-up was performed at 40% of maximal inspiratory pressure (MIP). Each protocol consisted of two sets of 30 repetitions (Marostegan et al., 2022; Demirkan et al., 2025).
  Arms: Athletic Warm-up Only; Inspiratory Warm-Up 40% MIP
Other: Sham — In addition to athletic warm-up an athletic warm-up protocol, participants performed inspiratory muscle warm-up (IMW) using the POWERbreathe® Plus Blue Medium Resistance (POWERbreathe International Ltd., Warwickshire, England UK). In the sham arm, inspiratory muscle warm-up was performed at 15% of maximal inspiratory pressure (MIP). Each protocol consisted of two sets of 30 repetitions (Marostegan et al., 2022; Demirkan et al., 2025).
  Arms: Athletic Warm-up Only; IW-SHAM

SUMMARY:
A single-blind, randomized crossover design was employed in this study. Two days before the study commenced, all participants were provided with detailed information about the warm-up protocols and tests to be conducted. Participants were brought to the standardized 400m-track for measurements a total of four times, with one-week intervals, beginning two days after the initial familiarization and information session. They were required not to perform any strenuous training and avoid long travels during 24 hours before the testing sessions. They were told to abstain from food intake for 3 hours before the protocol and avoid alcohol and caffeine for at least 24 hours prior to testing to ensure controlled conditions. The participants underwent four different warm-up protocols in a randomized order: one consisting of an athletic warm-up alone and three incorporating an inspiratory muscle warm-up at varying intensities in addition to the athletic warm-up. All warm-up protocols were administered one week apart, on the same day of the microcycle and at the same time, under relevant supervision. Various measurements were conducted at specific time points to assess physiological responses within each warm-up protocol. Accordingly, MIP and maximal expiratory pressure (MEP) tests were performed at the following time points: pre-warm-up, post-warm-up (pre-run), post-400-meter sprint, and at 1, 3, and 5 minutes after the run to evaluate inspiratory and expiratory muscle strength. Additionally, the Peak Inspiratory Flow Rate (PIFR) test was performed to determine inspiratory flow rate, and the Inhaled Volume (IV) test was conducted to measure the volume of air inhaled during inspiration. To objectively assess the effects of the warm-up protocols on sprint intensity and the recovery process, blood lactate testing was conducted. Furthermore, to monitor cardiovascular responses, heart rate measurements were recorded before the run, immediately after the 400-meter sprint, and at 1, 3, and 5 minutes post-run.

DETAILED DESCRIPTION:
Thirteen male 400-meter sprinters were included in analysis The participants' best recorded times ranged between 49.71 seconds and 51.74 seconds (Mean: 50.78±0.65 s). The required sample size was determined using*Power software (version 3.1.9.6; Dusseldorf, Germany), with a significance level of α = 0.05, statistical power (1 - β) = 0.95, and an effect size of ƒ = 0.5 (ANOVA with repeated measures, within interaction, 4 measurements) and totaled 10 participants. Initially, 14 athletes were recruited with convenience sampling by direct contact with coaches and athletes. One athlete dropped out during the study and did not complete all the required measurements and was not included in further analyses. All the participants were highly-trained athletes specializing in 400-meter sprint competitions, training six days per week.

Participants who voluntarily agreed to participate in the study and met the inclusion criteria were included after completing the Informed Consent Form. Upon obtaining approval from the responsible researcher and research supervisor, the warm-up protocols and physiological tests outlined in the study were initiated. The four different warm-up protocols were implemented in a randomized order: athletic warm-up alone, athletic warm-up + 60% inspiratory muscle warm-up, athletic warm-up + 40% inspiratory muscle warm-up, and athletic warm-up + 15% sham (placebo) inspiratory muscle warm-up. Immediately following each warm-up protocol, participants performed a 400-meter sprint, after which the physiological tests were repeated. The athletes were blinded to the applied protocol.

Athletic Warm-Up Protocol (AW) The athletic warm-up (AWU) consisted of 15 minutes of low-intensity running (rate of perceived effort 2-4 on 1-10 Borg Scale), followed by dynamic stretching exercises targeting the upper and lower extremities. In the final phase, running drills were performed, including three progressively increasing sprint efforts over a distance of approximately 30 meters.

Inspiratory Muscle Warm-up Protocols In addition to AWU an athletic warm-up protocol, participants performed inspiratory muscle warm-up (IMW) using the POWERbreathe® Plus Blue Medium Resistance (POWERbreathe International Ltd., Warwickshire, England UK) device at varying intensities. The IMW protocol was implemented at three different intensity levels: IW60, IW40, and IWPL. In the IW60 condition, inspiratory muscle warm-up was performed at 60% of maximal inspiratory pressure (MIP), while in IW40 and IWPL conditions, the intensity was set at 40% and 15% of MIP, respectively, with the latter serving as the sham protocolplacebo condition. Each protocol consisted of two sets of 30 repetitions.

MeasurementsTest Protocols Inspiratory and Expiratory Muscle Strength Test Maximal inspiratory pressure represents the highest negative intrathoracic pressure generated during inspiration, while MEP refers to the highest positive intrathoracic pressure produced by expiratory muscles under static conditions. These physiological parameters are commonly used for the objective assessment of respiratory muscle strength. For measurements, the Micro Medical-Carefusion Micro RPM (MicroMedical/CareFusion, Kent, UK) device, a validated assessment tool with real-time monitoring capability, was used. To prevent air leaks, participants' noses were occluded using a nasal clip during testing. For MEP measurement, participants were instructed to inhale maximally up to total lung capacity and then perform a forceful expiration through the mouthpiece. For MIP measurement, participants were instructed to exhale fully to residual volume, immediately followed by a maximal inspiratory effort. Each test was repeated at least three times, and testing was concluded when the difference between repeated measurements did not exceed 20%. The highest value was recorded as the final result. Participants were encouraged to exert maximum effort during all tests. All measurements were performed with participants in a seated position, following standardized guidelines of American Thoracic Society/European Respiratory Society .

Peak Inspiratory Flow Rate and Inhaled Volume Test Peak Inspiratory Flow Rate (PIFR) is a method used to assess respiratory muscle strength and airway resistance by measuring the maximum airflow rate (L/min) achieved during inspiration. Inhaled Volume (IV) measures the total volume of air (L) inhaled in a single breath, serving as an indicator of respiratory muscle capacity and pulmonary ventilation efficiency. A portable POWERbreathe® K5 device (POWERbreathe International Ltd., Warwickshire, England UK) was used for both assessments. Testing was conducted with participants seated, their noses occluded with a nose clip. Participants were instructed to exhale fully to residual volume, followed by a forceful maximal inspiration lasting at least one second. Each test was repeated three times, and the highest recorded value was used for analysis. Measurements of PIFR and IV were obtained simultaneously using the device's single-breath test mode.

Blood Lactate Test Blood lactate levels were measured using a portable and validated analysis device, the Lactate Scout Sport (EKF Diagnostics, Germany). All measurements were conducted according to standardized protocols to ensure accuracy and reliability. Capillary blood sampling was performed from the fingertip. Before sample collection, the skin was first cleansed and sweat was removed using an alcohol-based antiseptic, followed by rinsing with water for additional cleaning. A single-use lancet was then used to puncture the fingertip, and the first drop of blood was discarded. The subsequent drop was applied directly to the device's test strip for analysis. To prevent contamination and ensure measurement consistency, a different finger was used for each test. Additionally, the device's automatic calibration procedures were performed every 12 measurements.

Heat Rate A validated and highly accurate heart rate sensor (PolarPolar H10, Kempele, Finland) was used to measure heart rate, ensuring reliability and precision (Schaffarczyk et al., 2022) recorded in real time using the Polar Flow mobile application, which synchronizes wirelessly via Bluetooth with the sensor to provide instantaneous feedback on cardiac activity.

Determination of Sprint Time After completing the warm-up protocol, participants performed a 400-meter sprint test on a standard 400-meter outdoor tartan track (Lane 4) using their personal spiked running shoes previously used in competitions. The test was conducted using starting blocks, and at the beginning of each trial, a researcher with official sprint start officiating experience in track and field competitions gave the "Set" command. The sprint time was initiated automatically with the sound of a starting pistol connected to an optical sensor. Participants ran with maximum effort towards the finish line, where the time was stopped using optical sensors (DK-386, Turkey). Performance was recorded automatically. Participants were instructed to perform as if they were in a competitive race, but no pacing or race strategy guidance was provided. Due to the frequency of post-run measurements, each test was conducted individually to ensure accurate data collection.

Statistical analysis The normality of the distribution was evaluated with the Shapiro-Wilk test and visual assessment. The basic results are reported as mean and standard deviation. The statistical effects for running performance were evaluated by regular analysis of variance. The effects for time and the interaction between time and warm-up protocol for all other variables were analyzed using analysis of variance for repeated-measures. Mauchly's Test of Sphericity and Greenhouse-Geisser correction were used to identify and correct for the violation of sphericity. To account for multiple testing, the post-hoc Holm correction was applied, ensuring a stringent control of type I error. Effect sizes were calculated using partial eta squared (ηp²) and omega squared (ω²). The following values were suggested as small (0.01), medium (0.06) or large (0.14) effect sizes. A significance level of p < 0.05 was applied. All statistical analyses were performed using the JASP Team statistical package JASP (Amsterdam, Netherlands, version 0.17.2).

ELIGIBILITY:
Inclusion Criteria:

Athletes included in the study had previous competition experience in 400-meter track events on national level, no history of respiratory diseases, were non-smokers, and had not experienced any sports injuries in the past five months. All the participants were healthy and medically cleared to take part in competitive track and field.

Exclusion Criteria:

The exclusion criteria were: using any ongoing medication or using performance-enhancing substances, and any acute or chronic illness.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Running performance | 4 weeks
  After completing the warm-up protocol, participants performed a 400-meter sprint test on a standard 400-meter outdoor tartan track (Lane 4) using their personal spiked running shoes previously used in competitions. The test was conducted using starting blocks, and at the beginning of each trial, a researcher with official sprint start officiating experience in track and field competitions gave the "Set" command. The sprint time was initiated automatically with the sound of a starting pistol connected to an optical sensor. Participants ran with maximum effort towards the finish line, where the time was stopped using optical sensors (DK-386, Turkey). Performance was recorded automatically. Participants were instructed to perform as if they were in a competitive race, but no pacing or race strategy guidance was provided. Due to the frequency of post-run measurements, each test was conducted individually to ensure accurate data collection.
Maximal Pressures | 4 weeks
  Maximal inspiratory pressure represents the highest negative intrathoracic pressure generated during inspiration, while MEP refers to the highest positive intrathoracic pressure produced by expiratory muscles under static conditions. These physiological parameters are commonly used for the objective assessment of respiratory muscle strength (Gómez-Albareda et al., 2023; Evans & Whitelaw, 2009). For measurements, the Micro Medical-Carefusion Micro RPM (MicroMedical/CareFusion, Kent, UK) device, a validated assessment tool with real-time monitoring capability, was used (Erail & Mayda, 2023). To prevent air leaks, participants' noses were occluded using a nasal clip during testing. All measurements were performed with participants in a seated position, following standardized guidelines (American Thoracic Society/European Respiratory Society, 2002).
Peak Inspiratory Flow Rate | 4 weeks
  Peak Inspiratory Flow Rate (PIFR) is a method used to assess respiratory muscle strength and airway resistance by measuring the maximum airflow rate (L/min) achieved during inspiration (Ghosh et al., 2017). A portable POWERbreathe® K5 device (POWERbreathe International Ltd., Warwickshire, England UK) was used. Testing was conducted with participants seated, their noses occluded with a nose clip (Kowalski & Klusiewicz, 2023). Participants were instructed to exhale fully to residual volume (RV), followed by a forceful maximal inspiration lasting at least one second. Each test was repeated three times, and the highest recorded value was used for analysis. Measurements of PIFR were obtained simultaneously using the device's single-breath test mode (Demirkan et al., 2025).
Peak Inspiratory Flow Rate | 4 weeks
  Peak Inspiratory Flow Rate (PIFR) is a method used to assess respiratory muscle strength and airway resistance by measuring the maximum airflow rate (L/min) achieved during inspiration (Ghosh et al., 2017). A portable POWERbreathe® K5 device (POWERbreathe International Ltd., Warwickshire, England UK) was used for both assessments. It was conducted with participants seated, their noses occluded with a nose clip (Kowalski & Klusiewicz, 2023). Participants were instructed to exhale fully to residual volume (RV), followed by a forceful maximal inspiration lasting at least one second. Each test was repeated three times, and the highest recorded value was used for analysis. Measurements of PIFR and IV were obtained simultaneously using the device's single-breath test mode (Demirkan et al., 2025).
Inhaled Volume | 4 weeks
  (IV) measures the total volume of air (L) inhaled in a single breath, serving as an indicator of respiratory muscle capacity and pulmonary ventilation efficiency (Krause-Sorio et al., 2021). A portable POWERbreathe® K5 device (POWERbreathe International Ltd., Warwickshire, England UK) was used for the assessment. Testing was conducted with participants seated, their noses occluded with a nose clip (Kowalski & Klusiewicz, 2023). Participants were instructed to exhale fully to residual volume (RV), followed by a forceful maximal inspiration lasting at least one second. Each test was repeated three times, and the highest recorded value was used for analysis. Measurements of IV were obtained simultaneously using the device's single-breath test mode (Demirkan et al., 2025).
Blood lactate | 4 weeks
  Blood lactate levels were measured using a portable and validated analysis device, the Lactate Scout Sport (EKF Diagnostics, Germany). All measurements were conducted according to standardized protocols to ensure accuracy and reliability. Capillary blood sampling was performed from the fingertip. Before sample collection, the skin was first cleansed and sweat was removed using an alcohol-based antiseptic, followed by rinsing with water for additional cleaning. A single-use lancet was then used to puncture the fingertip, and the first drop of blood was discarded. The subsequent drop was applied directly to the device's test strip for analysis (Zhong et al., 2025). To prevent contamination and ensure measurement consistency, a different finger was used for each test. Additionally, the device's automatic calibration procedures were performed every 12 measurements.
Heart rate | 4 weeks
  A validated and highly accurate heart rate sensor (PolarPolar H10, Kempele, Finland) was used to measure heart rate, ensuring reliability and precision (Schaffarczyk et al., 2022). Heart rate data were continuously monitored and recorded in real time using the Polar Flow mobile application, which synchronizes wirelessly via Bluetooth with the sensor to provide instantaneous feedback on cardiac activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sport Sciences, Hitit University., Çorum, Corum Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The individual data of athletes will not be shared to protect their privacy and prevent any risk of identification. Maintaining confidentiality is essential to ensure that personal and performance-related information remains secure and is not misused. Small and elite athlete sample makes identification of the participants easy, based on their age, personal bests, and antrhopometric data. Therefore, only aggregated or anonymized data may be disclosed for research or reporting purposes, ensuring that no specific athlete can be identified from the information provided.